CLINICAL TRIAL: NCT00705159
Title: Safety and Efficacy of Zylet vs Lotemax, Tobramycin and Vehicle in Pediatric Blepharoconjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 550
Record Dates: First submitted 2008-06-20; First posted 2008-06-25 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Conjunctivitis
Keywords: Blepharokeratoconjunctivitis
MeSH Terms: conditions — Conjunctivitis | interventions — Loteprednol Etabonate; Tobramycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Loteprednol etabonate and tobramycin (Experimental): Drug: Zylet (loteprednol etabonate and tobramycin)
  Interventions: Drug: loteprednol etabonate and tobramycin
- Loteprednol etabonate (Active Comparator): Drug: Lotemax (loteprednol etabonate)
  Interventions: Drug: loteprednol etabonate
- Tobramycin (Active Comparator): Drug: Tobramycin
  Interventions: Drug: Tobramycin
- Vehicle (Placebo Comparator): Vehicle of Zylet
  Interventions: Drug: Vehicle of Zylet

INTERVENTIONS:
Drug: loteprednol etabonate and tobramycin — Topical ocular administration of loteprednol etabonate and tobramycin 4 times per day (QID) for 14 days.
  Other Names: Zylet
  Arms: Loteprednol etabonate and tobramycin
Drug: loteprednol etabonate — Topical ocular administration of Lotemax (loteprednol etabonate) QID for 14 days.
  Other Names: Lotemax
  Arms: Loteprednol etabonate
Drug: Tobramycin — Topical ocular administration of Tobramycin QID for 14 days.
  Arms: Tobramycin
Drug: Vehicle of Zylet — Topical ocular administration of the vehicle of Zylet QID for 14 days.
  Arms: Vehicle

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of Zylet in comparison with Lotemax, Tobramycin and the vehicle of Zylet for the treatment of blepharoconjunctivitis in pediatric subjects.

ELIGIBILITY:
Inclusion Criteria:

* children 0-6 years of age.
* clinical diagnosis of blepharoconjunctivitis
* Parent/guardian must understand, be willing and able to comply with all treatment and follow-up procedures.
* Parent/guardian must understand, be willing and able to provide informed consent and Health Insurance Portability Accountability Act (HIPAA) authorization.

Exclusion Criteria:

* Known hypersensitivity to corticosteroids, aminoglycosides, or any component of the study medication.
* Subjects who have a history of ocular surgery, including laser procedures, within the past 6 months.
* Subjects who are monocular.
* Subjects who have a history of any severe/serious ocular pathology or medical condition that could result in the subject's inability to complete the study.
* Subjects who have participated in an ophthalmic drug or device research study within 30 days prior to entry in this study.

Ages: 1 Week to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Ophthalmology of Erie, Erie, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 17 sites in the United States. First participant was enrolled on 6/26/2008 and last participant visit was 3/24/2010.
Pre-assignment Details: A total of 137 pediatric subjects, 0 to 6 years of age, of either gender and any race, who had a clinical diagnosis of blepharoconjunctivitis in at least one eye were randomized in this study. 126 Participants completed the study.
Groups:
- Loteprednol Etabonate and Tobramycin: Drug: Zylet (loteprednol etabonate 0.5% and tobramycin 0.3%)one or two drops in the study eye four times a day (QID).
- Loteprednol Etabonate: Drug: Lotemax (loteprednol etabonate 0.5%). One or two drops in study eye four times a day (QID).
- Tobramycin: Drug: Tobramycin 0.3%. One or two drops in study eye four times a day (QID).
- Vehicle: Vehicle of Zylet. One or two drops in study eye four times a day (QID).
Period: Overall Study
Arm/Group | Loteprednol Etabonate and Tobramycin | Loteprednol Etabonate | Tobramycin | Vehicle
Started | 34 | 35 | 34 | 34
Completed | 34 | 33 | 29 | 30
Not Completed | 0 | 2 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2
Not completed — Screen Failure | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol Etabonate and Tobramycin | Loteprednol Etabonate | Tobramycin | Vehicle | Total
Number analyzed (Participants) | 34 | 35 | 34 | 34 | 137
Age, Customized [Number; unit: participants]
  0-6 years | 34 | 35 | 34 | 34 | 137
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 15 | 14 | 57
  Male | 24 | 17 | 19 | 20 | 80
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 34 | 34 | 137

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Blepharoconjunctivitis Grade.
Description: Change from baseline to visit 4 in the total blepharoconjunctivitis grade. Graded on a scale of 0-4, 0 (none), 1 (minimal/trace), 2 (mild), 3 (moderate), and 4 (severe). Grade range from 0-32.
Time Frame: Baseline to 15 days
Population: Study eye, ITT Population, Non-missing data
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Loteprednol Etabonate and Tobramycin | Loteprednol Etabonate | Tobramycin | Vehicle
Number analyzed (Participants) | 34 | 35 | 34 | 33
Score on a scale | -11.41 (3.29) | -11.23 (3.98) | -10.68 (4.71) | -10.30 (5.19)

2. Secondary Outcome: Change From Baseline in Total Blepharoconjunctivitis Graded at Visit 2
Description: Change from baseline in total blepharoconjunctivitis grade to visit 2(day 3) measured on a scale of 0-4. 0 (none), 1 (minimal/trace), 2 (mild), 3 (moderate), and 4 (severe). Grade range from 0-32.
Time Frame: Baseline to Day 3
Population: Study eye, ITT population, non-missing data
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Loteprednol Etabonate and Tobramycin | Loteprednol Etabonate | Tobramycin | Vehicle
Number analyzed (Participants) | 34 | 34 | 32 | 31
Score on a scale | -7.32 (3.27) | -7.74 (3.90) | -5.94 (4.00) | -6.58 (3.46)

3. Secondary Outcome: Change From Baseline in Total Blepharoconjunctivitis Graded at Visit 3
Description: Change from baseline in total blepharoconjunctivitis grade to visit 3(day 7) measured on a scale of 0-4. 0 (none), 1 (minimal/trace), 2 (mild), 3 (moderate), and 4 (severe). Grade range from 0-32.
Time Frame: Baseline to Day 7
Population: Study eye ITT population, subjects with non-missing data
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Loteprednol Etabonate and Tobramycin | Loteprednol Etabonate | Tobramycin | Vehicle
Number analyzed (Participants) | 34 | 34 | 30 | 30
Score on a scale | -11.03 (3.20) | -10.94 (4.69) | -9.90 (3.80) | -10.03 (4.63)

ADVERSE EVENTS:
Time Frame: 15 days
Description: Safety population
Arm/Group | Loteprednol Etabonate and Tobramycin | Loteprednol Etabonate | Tobramycin | Vehicle
Serious Adverse Events (participants affected / at risk) | 2/34 | 2/35 | 2/34 | 1/33
Other Adverse Events (participants affected / at risk) | 2/34 | 2/35 | 2/34 | 2/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate and Tobramycin (N=34) | Loteprednol Etabonate (N=35) | Tobramycin (N=34) | Vehicle (N=33)
Respiratory distress (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) — Severe respiratory distress with moderate otitis media, unrelated to study drug or participation but due to concurrent illness.
Bronchiolitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (2) | 1 (2) — Bronchiolitis and dehydration unrelated to study drug or participation but due to concurrent illness.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate and Tobramycin (N=34) | Loteprednol Etabonate (N=35) | Tobramycin (N=34) | Vehicle (N=33)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) — Non-ocular AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.